CLINICAL TRIAL: NCT02686216
Title: Biodistribution, Pharmacokinetics, and Safety of F-18 THK-5351 PET in Alzheimer's Disease Patients and Healthy Subjects
Brief Title: Biodistribution, Pharmacokinetics, and Safety of F-18 THK-5351 PET in Alzheimer's Disease Patients and Healthy Subjects.(Positron Emission Tomograph )
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 104-2710A
Record Dates: First submitted 2016-01-15; First posted 2016-02-19 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2016-11

CONDITIONS: Alzheimer's Disease
Keywords: F-18 THK-5351 PET
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- F-18 THK-5351 (Experimental): F-18 THK-5351 imaging
  Interventions: Drug: F-18 THK-5351

INTERVENTIONS:
Drug: F-18 THK-5351 — Totally 24 subjects age 20-90 including 12 healthy cognitively intact subjects and 12 probably AD patients with NINCDS-ADRDA criteria. For disease subjects, caregiver should be able to report activities of daily living and their mental status. Patient should be able to give informed consent or have a caregiver give consent with subject assent.

SUMMARY:
Biodistribution, pharmacokinetics, and safety of F-18 THK-5351 PET in Alzheimer's disease patients and healthy subjects.

DETAILED DESCRIPTION:
Totally 24 subjects age 20-90 including 12 healthy cognitively intact subjects and 12 probably Alzheimer's dementia patients with NINCDS-ADRDA criteria. For disease subjects, caregiver should be able to report activities of daily living and their mental status. Patient should be able to give informed consent or have a caregiver give consent with subject assent.

ELIGIBILITY:
Healthy Inclusion Criteria:

* Neurologic testing. (MMSE 24-30, Wechsler Logical Memory score >5).
* Subjects must provide written inform consent.

Patients with AD Inclusion Criteria:

* Diagnosis of AD according to the clinical diagnostic criteria of "possible AD" with NINCDS-ADRDA criteria
* MMSE 20-26, Clinical dementia rating 0.5 or 1, Wechsler Logical Memory score<=4
* Patient who provide a written informed consent prior to study entry. (If the patient is incapable informed consent, the caregiver may consent on behalf of the patient. The caregiver should be able to report activities of daily living and their mental status.)

Exclusion Criteria:

* Pregnant or become pregnant
* Current breast feeding
* Clinically significant abnormal laboratory values
* Unstable medical or psychiatric illness.
* Cardiovascular disease (cardiac surgery or myocardial infarction within the last 6 months; unstable angina; decompensated congestive heart failure; significant cardiac arrhythmia; congenital heart disease).
* History of drug or alcohol abuse within the last year, or prior prolonged history of abuse. --History of severe allergic or anaphylactic reactions particularly to the tested drugs .
* PI assessment with high risk.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are to evaluate the dosimetry of novel radiotracer F-18 THK-5351 in human. | One year
  Time-integrated activity in each organ will be calculated by trapezoidal integration of the first 45 min of the organ's time-activity curve, followed by a single-exponential fit to the remaining data points (based on the 4 whole-body images) extrapolate to infinity, all base on non-decay-corrected data.Residence times will be obtained by dividing the time-integrated activity by the injected amount of activity.

SECONDARY OUTCOMES:
Optimal scanning time for brain imaging using F-18 THK-5351. | One year
  PET data will be acquired using SIMENS PET/CT or PET/MRI scanner with an axial field of view of 15.7cm. For PET/CT protocol, a 50-min dynamic brain PET scan (6x10s, 4x60s, 5x180s, 6x300s) will be started simultaneously with the injection of 10mCi of F-18 THK-5351 after a low-dose CT scan for patient positioning and attenuation correction.

REFERENCES:
- [Derived] Hsiao IT, Lin KJ, Huang KL, Huang CC, Chen HS, Wey SP, Yen TC, Okamura N, Hsu JL. Biodistribution and Radiation Dosimetry for the Tau Tracer 18F-THK-5351 in Healthy Human Subjects. J Nucl Med. 2017 Sep;58(9):1498-1503. doi: 10.2967/jnumed.116.189126. Epub 2017 Mar 23. PMID 28336780